CLINICAL TRIAL: NCT05884645
Title: The DAnish VIdeo IntubaTION (DA-VITION) Study: a Prospective Observational Cohort Study
Brief Title: The DAnish VIdeo IntubaTION (DA-VITION) Study
Acronym: DA-VITION
Status: Recruiting | Type: Observational
Sponsor: Lise Aunsholt (Other)
Collaborators: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Sponsor-Investigator, Lise Aunsholt, Associate Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: The DA-VITION study
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intubation Complication; Intubation; Difficult or Failed
Keywords: video-guided endotracheal intubation; artificial intelligence; videolaryngoscope

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing endotracheal intubation: Patients across all ages undergoing endotracheal intubation.
  Interventions: Procedure: Video-directed endotracheal intubation

INTERVENTIONS:
Procedure: Video-directed endotracheal intubation — There will be no intervention in this prospective observational cohort study. Endotracheal intubation is already used to secure the airway by placing an endotracheal tube into the trachea via the oral or nasal route. Indications include the need for airway control during general anaesthesia, mechanical ventilation, resuscitation, and various forms of acute respiratory distress.

SUMMARY:
This study aims to train an AI for video-directed endotracheal intubation (VITION) to recognise the anatomical structures of the upper airway during video-directed endotracheal intubations.

DETAILED DESCRIPTION:
Study design

The VITION study protocol describes the design of a prospective, observational study. Inclusion will commence in 2023 at the anesthesia and intensive care departments in the Capital Region of Denmark.

Participants

Patients across all ages are eligible for inclusion if they are undergoing video-directed oral or nasal endotracheal intubation.

Exclusion criteria

Patients are excluded if they adhere to one of the exclusion criteria:

* Upper airway malformations (e.g., laryngomalacia, vocal cord paralysis, and subglottic stenosis17,18).
* Failed attempt by video laryngoscopy due to malfunctioning equipment.
* Missing or corrupted video recording.
* Informed consent is not obtained from the participants or participants' parents / legal guardians.

Interventions and comparisons

This prospective, observational study will have no interventions or comparisons.

Primary objective

The primary objective is to characterize anatomical landmarks and performances of intubations in a large and diverse pool of clinicians and patients.

ELIGIBILITY:
Patients are eligible if they adhere to all the following inclusion criteria:

● Undergoing video-directed oral or nasal endotracheal intubation.

Exclusion criteria

Patients are excluded if they adhere to one of the exclusion criteria:

* Upper airway malformations (e.g., laryngomalacia, vocal cord paralysis, and subglottic stenosis).
* Failed attempt by video laryngoscopy due to malfunctioning equipment.
* Missing or corrupted video recording.
* Informed consent is not obtained from the participants or participants' parents / legal guardians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will include patients across all ages are eligible for inclusion if they are undergoing video-directed oral or nasal endotracheal intubation in the Capital Region of Denmark.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the AI algorithm to recognise the anatomical landmarks in the upper airway. | The landmarks will be identified on the multimedia file from the procedure.
  Accuracy of the AI algorithm to recognise the anatomical landmarks in the upper airway.
Sensitivity of the AI algorithm to recognise the anatomical landmarks in the upper airway. | The landmarks will be identified on the multimedia file from the procedure.
  Sensitivity of the AI algorithm to recognise the anatomical landmarks in the upper airway.
Specificity of the AI algorithm to recognise the anatomical landmarks in the upper airway. | The landmarks will be identified on the multimedia file from the procedure.
  Specificity of the AI algorithm to recognise the anatomical landmarks in the upper airway.
AUC of the AI algorithm to recognise the anatomical landmarks in the upper airway. | The landmarks will be identified on the multimedia file from the procedure.
  AUC of the AI algorithm to recognise the anatomical landmarks in the upper airway.

SECONDARY OUTCOMES:
Time consumption of the course. | During the procedure.
  A course is defined as one method for intubation (i.e., the same airway device, approach, and medication regimen). Many attempts by multiple providers are allowed within a given course as long as all attempts are made using the same method.
Number of attempts. | During the procedure.
  The number of attempts (one, two, and three or more).
Successful endotracheal intubation. | During the procedure.
  Successful endotracheal intubation is defined as correct endotracheal tube placement in the trachea confirmed by chest rise, auscultation, waveform monitor for end-tidal CO2, and/or chest radiograph in first, second, or three attempts.10,19 First-attempt success is defined according to previous studies as successful intubation on the first attempt by the first provider. Success within two attempts is defined as successful intubation on the second attempt by the same provider. Success within 3 attempts is defined as successful intubation on any attempt by the same provider.
Overall course success. | During the procedure.
  Overall course success is defined as successful intubation by any provider on any attempt within that course.
Severe oxygen desaturations | During the procedure.
  Severe oxygen desaturations are defined according to previous studies as a 20% or more decrease in oxygen saturation from the highest level immediately before the first attempt.
Non-severe TIAEs | 72 hours after the procedure
  Non-severe TIAEs: Oesophageal intubation with immediate recognition, dysrhythmia including any duration of heart rate <60 beats per minute without chest compressions, main-stem bronchial intubation, emesis without aspiration, pain or agitation requiring additional medications causing a delay in intubation, epistaxis, lip trauma, dental injury, medication error, and hypertension.
Severe TIAEs | 72 hours after the procedure
  Severe TIAEs: Cardiac arrest requiring chest compressions, oesophageal intubation with delayed recognition (defined as placement of the endotracheal tube into the oesophagus or hypopharynx with clinical deterioration, e.g., desaturation, before removal of the misplaced tube), emesis with aspiration, hypotension requiring therapy, laryngospasm, pneumothorax or pneumo-mediastinum, and direct airway injury (e.g., vocal cord injury, laryngeal injury, tracheal injury, false passage creation).

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Breindahl, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Capital Region of Denmark, Copenhagen

IPD SHARING:
Plan to Share IPD: No
The Capital Region in Denmark retains all rights to the collected data, which must not be shared without approval.